CLINICAL TRIAL: NCT03877978
Title: Evaluation of the Incidence of Acute Kidney Attack by Dosing Nephrocheck® in Severe Traumatized Patients
Brief Title: Acute Kidney Attack in Severe Traumatized Patients
Acronym: NEPHROTRAUMA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0903
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe traumatized patients: Severe traumatized patients with an Index Severity Score (ISS) ≥ 15 admitted to the trauma center of Edouard Herriot Hospital.
  Interventions: Biological: Nephrocheck test

INTERVENTIONS:
Biological: Nephrocheck test — Nephrocheck® measurement on urine sample at different timepoints.

SUMMARY:
Acute Kidney Injury (AKI) is a common complication of severe traumatized patients. The diagnosis is often delayed. The Nephrocheck® test allows an earlier assessment of renal stress. The objective of our study is to determine the incidence of risk of AKI in severe traumatized patients within the first 24 hours after their admission to our trauma center. The risk of AKI is defined by a NephroCheck® test >0.3

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* trauma patients with ISS ≥15
* patient admitted to the resuscitation bay of Edouard Herriot Hospital

Exclusion Criteria:

* anuric patient
* opposition of the patient (or a trusted person) to participate
* pregnant or lactating woman
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe traumatized patients with an ISS ≥ 15 admitted to the trauma center of Edouard Herriot Hospital
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with Nephrocheck score > 0,3 | Up to 24 hours after trauma
  Incidence of severe traumatized patient at risk of AKI as defined by Nephrocheck test score > 0,3 within the first 24 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Violette Zorio, Principal Investigator — Intensive Care Unit, Pavillon H - Réanimation chirurgicale. Edouard Herriot hospital 5 place d'Arsonval - 69003 Lyon FRANCE
Locations (1):
- Hôpital Edouard Herriot, Lyon, France